CLINICAL TRIAL: NCT02370888
Title: A Phase I Clinical Trial to Evaluate the Maximally Tolerated Dose (MTD), Dose Limiting Toxicities (DLTs) and Safety Profiles of Increasing Doses of Lenalidomide After Allo-HCT in AML and MDS Subjects With Minimal Residual Disease (MRD) Detected by the CD34+ Mixed Chimerism Analysis (UF-BMT-MRD-101)
Brief Title: Lenalidomide After Allo-Hematopoietic Cell Transplant (HCT) in Acute Myelogenous Leukemia (AML) and Myelodysplastic Syndromes (MDS) Subjects With Minimal Residual Disease
Acronym: UF-BMT-MRD-101
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University of Florida (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WIRB20151509; RV-CL-AML-PI-002987 (Other Grant/Funding Number: Celgene Corporation)
Record Dates: First submitted 2015-02-10; First posted 2015-02-25 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Leukemia, Myeloid; Myelodysplastic Syndromes
Keywords: Lenalidomide; Hematopoietic Stem Cell Transplantation; Peripheral Blood Stem Cell Transplantation
MeSH Terms: conditions — Leukemia, Myeloid; Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lenalidomide (Experimental): Lenalidomide will be administered for a total of 42 days.
  The dose levels of lenalidomide will be as follows:
  * Dose Level 1: 2.5 mg PO QOD Day 1-21 for 28-day cycle X 2 cycles
  * Dose Level 2: 2.5 mg PO QD Day 1-21 for 28-day cycle X 2 cycles
  * Dose Level 3: 5 mg PO QD Day 1-21 for 28-day cycle X 2 cycles
  * Dose Level 4: 7.5 mg PO QD Day 1-21 for 28-day cycle X 2 cycles
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Subjects will be enrolled in cohorts of three (3). Lenalidomide will be administered for 21 consecutive days in a 28 day cycle X 2 cycles. The starting dose will be 2.5 mg given orally every other day for 21 days.
  Other Names: Revlimid

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose, dose limiting side effects, and the safety of increasing doses of lenalidomide in patients with AML and MDS who have a small amount of detectable disease after allogeneic stem cell transplant.

DETAILED DESCRIPTION:
All subjects entering the screening phase will receive a unique subject number. This number will be used to identify the subject throughout the study. Additional test to include: physical examinations, blood tests, and if applicable pregnancy test will be performed as part of participation in this research study.

Lenalidomide will be administered for a total of 42 days. The starting dose will be 2.5 mg given orally every other day on days 1-21 of a 28-day cycle for 2 cycles. Dose escalations and de-escalations will be made until the maximum tolerated dose is reached.

The dose levels of lenalidomide will be as follows:

Dose Level 1: 2.5 mg

Dose Level 2: 2.5 mg

Dose Level 3: 5 mg

Dose Level 4: 7.5 mg

Doses should be taken at approximately the same time each day.

Subjects must be instructed to swallow lenalidomide capsules whole with water at the same time each day. Do not break, chew or open the capsules.

Each subject will keep an accurate record of lenalidomide dosing on the Subject Dosing Diary. This diary will be kept in the research record as source documentation of lenalidomide dosing. Study personnel will review the dosing instructions with each subject at each study visit. Subjects will be asked to bring any unused drug and empty drug containers to the study site at the next visit for reconciliation with the Subject Dosing Diary.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age;
2. Subjects must be post-allogeneic transplant from any donor source;
3. Subjects must have either:

   1. High risk CD34+ AML (de novo or secondary, and any WHO 2008 classification excluding acute promyelocytic leukemia). High risk AML is defined as (a) disease status beyond complete remission (CR) #1 at transplant or (b) treatment related AML or (c) presence of adverse cytogenetics including inv(3); t(3;3); t(6;9); t(v;11); -5 or del(5q); -7; abnl(17p) or complex karyotype; or
   2. High risk CD34+ MDS (WHO 2008 classification). High risk is defined as (a) blast count ≥5% at the time of transplant or (b) treatment related MD or (c) presence of adverse cytogenetics including -7/del7q or complex karyotype;
4. For AML subjects, they must have a documented CR within 45 days prior to allo-HCT;
5. For MDS subjects, they must have < 20% myeloblasts in the bone marrow within 45 days prior to allo-HCT;
6. Subject Karnofsky performance status must be ≥ 70;
7. Subjects must be platelet transfusion independent (Platelet transfusion independence is defined as 7 days or greater without a platelet transfusion);
8. Neutrophil count ≥ 1.0 thou/mm3 and platelet count ≥ 30 thou/mm3;
9. Subjects must have total bilirubin ≤ 2 mg/dL;
10. Subjects must have serum AST and ALT levels ≤ 2.5 times upper limit of normal;
11. Subjects must have serum creatinine < 2.5 times upper limit of normal and a calculated creatinine clearance > 30 ml/min by Cockcroft-Gault formula (see Appendix I: Cockcroft-Gault Creatinine Clearance Calculation);
12. All study participants who will receive lenalidomide based on the CD34+ chimerism testing must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of the REMS® program;
13. Females of child-bearing potential (i.e., women who are premenopausal or not surgically sterile) may participate, provided they meet the following conditions:

    a) Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program; and
14. Written, voluntary informed consent, willingness, and ability to comply with all study procedures.

Exclusion Criteria:

1. CD34- AML or MDS;
2. Inability to give informed consent;
3. Uncontrolled active infection(s) requiring intravenous antibiotics;
4. Known or suspected hypersensitivity to lenalidomide;
5. Grade II-IV acute GVHD or extensive GVHD;
6. Not able to swallow the lenalidomide capsule as a whole;
7. Female subjects who are pregnant or nursing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxim N. Norkin, M.D., Ph.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida Shands Cancer Center, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, enrollment is completion of informed consent. 11 subjects were enrolled- 2 did not meet eligibility and 9 did. Of the 9 eligible subjects- 3 received protocol treatment assignment, 5 did not have their chimerism drop, per protocol, below 90% at day 60 or 90 post-transplant, and 1 withdrew consent prior to assignment.
Groups:
- Dose Escalation of Lenalidomide: Participants in the Arm only received Dose Level 1: 2.5 mg PO QOD Day 1-21 for 28-day cycle X 2 cycles
Period: Overall Study
Arm/Group | Dose Escalation of Lenalidomide
Started | 9
Proceed to Treatment | 3
Completed | 1
Not Completed | 8
Not completed — disease progression | 2
Not completed — did not meet chimerism criteria | 6

BASELINE CHARACTERISTICS:
Population: Subsequent cohort requirements for analysis not met.
Groups:
- Dose Level 1: 2.5 mg PO QOD Day 1-21 for 28 day cycle X 2 Enrolled 3 subjects
- Dose Level 2: 2.5 mg PO QD Day 1-21 for 28 day cycle X 2 cycles
- Dose Level 3: 5 mg PO QD Day 1-21 for 28 day cycle X 2 cycles
- Dose Level 4: 7.5 mg PO QD Day 1-21 for 28 day cycle X 2 cycles
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Total
Number analyzed (Participants) | 3 | 0 | 0 | 0 | 3
Age, Customized [Count of Participants; unit: Participants] | 3 |  |  |  | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Gender: Female | 1 |  |  |  | 1
  Gender: Male | 2 |  |  |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  |  |  | 0
  Not Hispanic or Latino | 3 |  |  |  | 3
  Unknown or Not Reported | 0 |  |  |  | 0
Number of Participants with CD34 donor chimerism drop [Count of Participants; unit: Participants] — The number of study participants who experienced a CD34+ donor chimerism drop of less than or equal to 90% in allo-hematopoietic stem cell transplantation patients. CD34+ chimerism measurement is obtained via a peripheral blood draw.
  Participants | 3 |  |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Lenalidomide
Description: To determine safety and the maximum tolerated dose of lenalidomide after allo-HCT in AML and MDS subjects with MRD detected by the CD34+ mixed chimerism analysis.
Time Frame: Up to 72 days
Population: Cohort requirements for analysis not met. MTD could not be assessed as only a single dose level was tested. No dose escalation was performed.
Groups:
- Dose Level 1: Lenalidomide 2.5 mg by mouth every other day for twenty-one days of a 28 day cycle for 2 cycles.
Arm/Group | Dose Level 1
Number analyzed (Participants) | 0

2. Secondary Outcome: CD34+ Mixed Chimerism
Description: To monitor changes in the CD34+ mixed chimerism after allo-HCT in AML and MDS subjects with detectable MRD in response to escalating doses of lenalidomide.
Time Frame: Up to 120 days
Population: No participant met the requirements for the efficacy population (at least 21 days of the study drug and at least one post-cycle efficacy assessment). Therefore, no data were collected for this assessment.
Groups:
- Dose Level 1: Lenalidomide 2.5 mg by mouth every other day for twenty-one days of a 28 day cycle for two cycles.
- Dose Level 2: Lenalidomide 2.5 mg by mouth daily for twenty-one days of a 28 day cycle for two cycles.
- Dose Level 3: Lenalidomide 5 mg by mouth daily for twenty-one days of a 28 day cycle for 2 cycles.
- Dose Level 4: Lenalidomide 7.5 mg by mouth daily for twenty-one days of a 28 day cycle for 2 cycles.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Dose Level 1: 2.5 mg PO QOD Day 1-21 for 28 Day Cycle X 2: Subjects will be enrolled in cohorts of three (3). Lenalidomide will be administered for 21 consecutive days in a 28 day cycle X 2 cycles.
Arm/Group | Dose Level 1: 2.5 mg PO QOD Day 1-21 for 28 Day Cycle X 2
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 2.5 mg PO QOD Day 1-21 for 28 Day Cycle X 2 (N=3)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2)
General disorders and administration site conditions (General disorders) | 2 (4)
Investigations (Investigations) | 2 (18)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (5)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (10)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (5)
Infections and infestations (Infections and infestations) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/88/NCT02370888/Prot_SAP_000.pdf